CLINICAL TRIAL: NCT00440011
Title: Bimatoprost 0.03% Versus Travoprost 0.004% in Patients Currently on Latanoprost 0.005%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Medical Affairs Director, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MA-LUM01
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Results first posted 2008-09-26 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Bimatoprost; Ophthalmic Solutions; Travoprost

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bimatoprost 0.03% eye drops
- 2 (Active Comparator)
  Interventions: Drug: travoprost 0.004% eye drops

INTERVENTIONS:
Drug: bimatoprost 0.03% eye drops — bimatoprost 0.03% 1 drop nightly for 3 months
  Other Names: Lumigan®
  Arms: 1
Drug: travoprost 0.004% eye drops — travoprost 0.004% 1 drop nightly for 3 months
  Other Names: Travatan®
  Arms: 2

SUMMARY:
Patients with glaucoma or ocular hypertension currently being treated with latanoprost 0.005%, and in need of additional IOP lowering, will be randomized to receive either bimatoprost 0.03% or travoprost 0.004% in place of latanoprost 0.005%

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma or ocular hypertension in both eyes
* Currently being treated with latanoprost 0.005% daily and in need of additional IOP-lowering
* Best-corrected visual acuity of 20/100 or better in each eye
* Visual field within 6 months of study entry

Exclusion Criteria:

* Secondary glaucoma
* Active intraocular inflammation or macular edema
* Intraocular surgery or laser surgery within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2006-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Allergan
Locations (1):
- San Diego, California, United States

REFERENCES:
- [Background] Kammer JA, Katzman B, Ackerman SL, Hollander DA. Efficacy and tolerability of bimatoprost versus travoprost in patients previously on latanoprost: a 3-month, randomised, masked-evaluator, multicentre study. Br J Ophthalmol. 2010 Jan;94(1):74-9. doi: 10.1136/bjo.2009.158071. Epub 2009 Sep 1. PMID 19726422

RESULTS

PARTICIPANT FLOW:
Groups:
- Bimatoprost: bimatoprost 0.03% 1 drop nightly for 3 months
- Travoprost: travoprost 0.004% 1 drop nightly for 3 months
Period: Overall Study
Arm/Group | Bimatoprost | Travoprost
Started | 131 | 135
Completed | 127 | 132
Not Completed | 4 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost | Travoprost | Total
Number analyzed (Participants) | 131 | 135 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (12.3) | 62.7 (12.4) | 63.0 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 66 | 147
  Male | 50 | 69 | 119
Region of Enrollment [Number; unit: participants]
  United States | 131 | 135 | 266

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: Intraocular Pressure
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Bimatoprost | Travoprost
Number analyzed (Participants) | 127 | 132
mm Hg | 17 (3.1) | 17.5 (2.6)
Statistical Analysis 1: Comparison: Bimatoprost vs Travoprost; Test type: Superiority or Other; p = 0.024, ANCOVA

2. Secondary Outcome: Tolerability - Conjunctival Hyperemia
Description: Conjunctival Hyperemia: Number of participants with at least 1 grade increase in severity from baseline. A five grade scale from 0 to 3 (0 = none, +0.5 = trace, 1 = mild, 2 = moderate, 3 = severe)
Time Frame: Month 3
Measure: Number; unit: participants
Arm/Group | Bimatoprost | Travoprost
Number analyzed (Participants) | 127 | 132
participants | 15 | 22

ADVERSE EVENTS:
Arm/Group | Bimatoprost | Travoprost
Serious Adverse Events (participants affected / at risk) | 1/131 | 0/133
Other Adverse Events (participants affected / at risk) | 21/131 | 22/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost (N=131) | Travoprost (N=133)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost (N=131) | Travoprost (N=133)
Ocular Hyperaemia (Eye disorders) | 4 | 1
Eye Pruritus (Eye disorders) | 3 | 1
Conjunctival Hyperaemia (Eye disorders) | 1 | 2
Punctate keratitis (Eye disorders) | 1 | 2
Eye Irritation (Eye disorders) | 2 | 0
Growth of Eyelashes (Eye disorders) | 2 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 2
Abnormal Sensation in Eye (Eye disorders) | 1 | 0
Eye Discharge (Eye disorders) | 1 | 0
Eyelid Margin Crusting (Eye disorders) | 0 | 1
Lenticular Opacities (Eye disorders) | 0 | 1
Instillation Site Pruritus (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Sensation of Foreign Body (General disorders) | 0 | 1
Conjunctivitis Viral (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Stomach Discomfort (Gastrointestinal disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1
Foreign Body in Eye (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hyperaemia (Vascular disorders) | 0 | 1
Blepharitis (Eye disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less